CLINICAL TRIAL: NCT04215029
Title: Reducing Prostate Cancer Disparities Among African Americans
Brief Title: Lifestyle Intervention for the Reduction of Prostate Cancer Disparities Among African Americans
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Brander Beacons Cancer Research (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-0361; NCI-2019-05912 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0361 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-11-26; First posted 2020-01-02 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Cancer Survivor; Partner; Spouse; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Interviews as Topic; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (exercise plan, coaching calls, nutrition counseling) (Experimental): Patients and their partners receive an exercise plan and printed materials that includes instructions for walking or other moderate-intensity activities. Patients and their partners also receive coaching calls discussing physical activity and diet related questions, each lasting 45-60 minutes and occurring every 2 weeks for 6 months. In addition, patients and their partners complete 2 nutrition counseling sessions over 1 hour each at baseline and before month 3 with an MD Anderson registered dietitian.
  Interventions: Behavioral: Exercise Intervention; Other: Informational Intervention; Other: Nutritional Assessment; Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention
- Group II (physical activity/healthy eating information) (Active Comparator): Patients and their partners receive information/materials regarding physical activity and healthy eating.
  Interventions: Other: Informational Intervention; Other: Questionnaire Administration
- Provider Interviews (interviews) (Experimental): Healthcare providers participate in an interview regarding their opinions on family-focused care and its ability to improve health behaviors.
  Interventions: Other: Interview

INTERVENTIONS:
Behavioral: Exercise Intervention — Receive exercise plan
  Arms: Group I (exercise plan, coaching calls, nutrition counseling)
Other: Informational Intervention — Receive printed exercise materials
  Arms: Group I (exercise plan, coaching calls, nutrition counseling)
Other: Informational Intervention — Receive physical activity and healthy eating information/materials
  Arms: Group II (physical activity/healthy eating information)
Other: Interview — Participate in interview
  Arms: Provider Interviews (interviews)
Other: Nutritional Assessment — Complete nutrition counseling sessions
  Other Names: Dietary Assessment; dietary counseling; nutritional counseling
  Arms: Group I (exercise plan, coaching calls, nutrition counseling)
Other: Questionnaire Administration — Ancillary studies
  Arms: Group I (exercise plan, coaching calls, nutrition counseling); Group II (physical activity/healthy eating information)
Behavioral: Telephone-Based Intervention — Receive coaching calls
  Arms: Group I (exercise plan, coaching calls, nutrition counseling)

SUMMARY:
This trial studies how well a lifestyle intervention works in reducing prostate cancer disparities among African American prostate cancer patients and their spouses or romantic partners. A lifestyle intervention may help researchers learn if social support can help African American prostate cancer patients and their partners improve their quality of life, support from their partner, physical activity, diet, and inflammation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To expand an existing couple-based behavioral intervention developed for African American (AA) or Hispanic men on active surveillance (Watchful Living; protocol #: 2017-0556) to AA prostate cancer (PCa) survivors who underwent active treatments to examine its feasibility of recruiting AA PCa survivor-partner dyads (N = 40 dyads) and implementing a lifestyle intervention.

SECONDARY OBJECTIVES:

I. Evaluate a preliminary efficacy of the intervention in improving quality of life, physical activity, nutrient intake, and inflammation.

II. Explore psychosocial mediators and moderators of the intervention. III. Conduct a process evaluation. IV. Assess healthcare-provider level factors (with N=15 providers) that influence both survivors' and partners' healthy lifestyle behaviors.

OUTLINE: Patients and their partners are randomized to 1 of 2 groups.

GROUP I: Patients and their partners receive an exercise plan and printed materials that includes instructions for walking or other moderate-intensity activities. Patients and their partners also receive coaching calls discussing physical activity and diet related questions, each lasting 45-60 minutes and occurring every 2 weeks for 6 months. In addition, patients and their partners complete 2 nutrition counseling sessions over 1 hour each at baseline and before month 3 with an MD Anderson registered dietitian.

GROUP II: Patients and their partners receive information/materials regarding physical activity and healthy eating.

PROVIDER INTERVIEWS: Healthcare providers participate in an interview regarding their opinions on family-focused care and its ability to improve health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible, prostate cancer survivors must self-identify as black or African American
* Prostate cancer survivors must have 0-III stage prostate cancer
* Prostate cancer survivors must have completed therapy (e.g., surgery, chemotherapy [chemo] and/or radiation)
* Prostate cancer survivors must enroll with a spouse or a romantic partner
* Prostate cancer survivors must not meet physical activity recommendation (i.e., 150 minutes of moderate intensity physical activity per week)
* Prostate cancer survivors must be willing and able to be physically active, as determined by responses to the Physical Activity Readiness Questionnaire (PAR-Q)
* Prostate cancer survivors must not participate in another physical activity, diet, or lifestyle program
* Prostate cancer survivors must have a valid home address and telephone number
* Prostate cancer survivors must be able to access internet over a smartphone or a computer at home or other location (e.g., work, church, library, community center, etc.)
* To be eligible, spouses or romantic partners must be >=18 years of age
* Spouses or romantic partners must enroll with a spouse or a romantic partner with prostate cancer
* Spouses or romantic partners must live together with the survivors
* Spouses or romantic partners must not have major health problems (e.g., cancer, dementia, stroke, and heart and lung diseases)
* Spouses or romantic partners must be willing and able to be physically active, as determined by responses to the Physical Activity Readiness Questionnaire (PAR-Q)
* To be eligible, healthcare providers must be currently providing care with individuals diagnosed with prostate cancer
* Any professionals such as surgical and medical oncologists, fellows, nurse practitioners, physical assistants, and primary care physicians will be eligible

Exclusion Criteria:

* Prostate cancer survivors will be excluded if they are not married or partnered
* Prostate cancer survivors will be excluded if they have an active noncutaneous malignancy at any site
* Prostate cancer survivors will be excluded if they had a prior history of other cancer or have metastatic cancer
* Prostate cancer survivors will be excluded if they have planned concomitant immunotherapy, hormonal therapy, chemotherapy, or radiation therapy during the study period
* Prostate cancer survivors will be excluded if they are on active surveillance
* Prostate cancer survivors will be excluded if they enrolled in a protocol #: 2017-0556
* Prostate cancer survivors will be excluded if they are not able to understand and speak English
* Spouses or romantic partners who are not able to understand and speak English will be excluded
* Also, spouses or romantic partners who enrolled in a protocol (#2017-0556) will be excluded
* There are no exclusion criteria for healthcare providers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Implementing a lifestyle intervention and active surveillance on couple-based behavioral intervention developed for African American (AA) or Hispanic men | up to 6 months
  We will calculate rates of recruitment and retention, along with 90% confidence intervals (CIs). Participant feedback will be summarized using means and standard deviations (SDs)

CONTACTS AND LOCATIONS:
Overall Officials: Dalnim Cho, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org